CLINICAL TRIAL: NCT03970096
Title: A Phase II Randomized Controlled Trial Comparing GVHD-Reduction Strategies for Allogeneic Peripheral Blood Transplantation (PBSCT) for Patients With Acute Leukemia or Myelodysplastic Syndrome: Selective Depletion of CD45RA+ Naïve T Cells (TND) vs. Post-Transplantation Cyclophosphamide (PTCy)
Brief Title: Graft Versus Host Disease-Reduction Strategies for Donor Blood Stem Cell Transplant Patients With Acute Leukemia or Myelodysplastic Syndrome (MDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1005364; 9749 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2019-03188 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
Keywords: Lymphoid Leukemia; Myeloid and Monocytic Leukemia; Other Hematopoietic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphoid; Leukemia, Monocytic, Acute | interventions — Whole-Body Irradiation; Thiotepa; fludarabine; Tacrolimus; Methotrexate; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Cyclosporins; Sirolimus; Busulfan; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A1 (TBI, TnD) (Experimental): Patients undergo TBI BID on days -10 to -7, and receive thiotepa IV over 3 hours on days -6 and -5, fludarabine IV over 30 to 60 minutes on days -6 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, CD34+ enriched CD45RA-depleted donor T-lymphocytes IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Radiation: Total-Body Irradiation; Drug: Thiotepa; Drug: Fludarabine; Drug: Tacrolimus; Biological: Allogeneic CD34+-enriched and CD45RA-depleted PBSCs; Drug: Methotrexate; Drug: Cyclosporine; Drug: Sirolimus; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection
- Arm A2 (busulfan, TnD) (Experimental): Patients receive fludarabine IV over 30 to 60 minutes on days -6 to -2, busulfan IV over 180 minutes on days -5 to -2, and undergo TBI BID on day -1. Patients also receive tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, CD34+ enriched CD45RA-depleted donor T-lymphocytes IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Drug: Fludarabine; Drug: Tacrolimus; Biological: Allogeneic CD34+-enriched and CD45RA-depleted PBSCs; Drug: Methotrexate; Drug: Cyclosporine; Drug: Sirolimus; Drug: Busulfan; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection
- Arm C1 (TBI, PTCy, tacrolimus) (Experimental): Patients undergo TBI BID on days -4 to -2 or -3 to -1, and receive PBSC IV on day 0. Patients also receive cyclophosphamide IV over 1 to 2 hours on days 3 and 4, and tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day 5. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Radiation: Total-Body Irradiation; Drug: Tacrolimus; Drug: Cyclophosphamide; Biological: Peripheral Blood Stem Cell; Drug: Cyclosporine; Drug: Sirolimus; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection
- Arm C2 (busulfan, PTCy, tacrolimus) (Experimental): Patients receive fludarabine IV over 30 to 60 minutes on days -5 to -2, busulfan IV over 180 minutes on days -5 to -2, PBSC IV on day 0, cyclophosphamide IV over 1 to 2 hours on days 3 and 4, and tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day 5. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Drug: Fludarabine; Drug: Tacrolimus; Drug: Cyclophosphamide; Biological: Peripheral Blood Stem Cell; Drug: Cyclosporine; Drug: Sirolimus; Drug: Busulfan; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection
- Arm D1 (TBI, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021] (Experimental): Patients undergo TBI BID on days -6 to -4, and receive cyclophosphamide IV over 1 hour on days -3 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, PBSC IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Radiation: Total-Body Irradiation; Drug: Tacrolimus; Drug: Methotrexate; Drug: Cyclophosphamide; Biological: Peripheral Blood Stem Cell; Drug: Cyclosporine; Drug: Sirolimus; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection
- Arm D2 (busulfan, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021] (Experimental): Patients receive busulfan IV over 180 minutes on days -8 to -5, cyclophosphamide IV over 1 hour on days -3 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, PBSC IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid). Patients also undergo bone marrow aspiration/biopsy, ECHO or MUGA scan, and collection of blood samples throughout the trial.
  Interventions: Drug: Tacrolimus; Drug: Methotrexate; Drug: Cyclophosphamide; Biological: Peripheral Blood Stem Cell; Drug: Cyclosporine; Drug: Sirolimus; Drug: Busulfan; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection

INTERVENTIONS:
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation; TBI; Whole Body Irradiation; SCT_TBI; Total-Body Irradiation Prior to Stem Cell Transplant
  Arms: Arm A1 (TBI, TnD); Arm C1 (TBI, PTCy, tacrolimus); Arm D1 (TBI, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]
Drug: Thiotepa — Given IV
  Other Names: Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Triethylene; Triethylenethiophosphoramide; SH-105
  Arms: Arm A1 (TBI, TnD)
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Arm A1 (TBI, TnD); Arm A2 (busulfan, TnD); Arm C2 (busulfan, PTCy, tacrolimus)
Drug: Tacrolimus — Given IV
  Other Names: Prograf; Protopic; FK-506
Biological: Allogeneic CD34+-enriched and CD45RA-depleted PBSCs — Given IV
  Other Names: Allogeneic TN-depleted CD34-preserved PBSCs; Allogeneic TND- CD34+ PBSCs; Donor-derived TN Cell Depleted CD34-enriched PBSCs; Naive T-cell Depleted CD34+ Allogeneic Peripheral Blood Stem Cells
  Arms: Arm A1 (TBI, TnD); Arm A2 (busulfan, TnD)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; Emthexat; Emtexate; Farmitrexat; Methotrexate LPF; Methylaminopterin; Methotrexatum; Metotrexato
  Arms: Arm A1 (TBI, TnD); Arm A2 (busulfan, TnD); Arm D1 (TBI, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]; Arm D2 (busulfan, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]
Drug: Cyclophosphamide — Given IV
  Other Names: Ciclofosfamida; Ciclofosfamide; Cicloxal; Claphene; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cytophosphan; Asta B 518; WR-138719
  Arms: Arm C1 (TBI, PTCy, tacrolimus); Arm C2 (busulfan, PTCy, tacrolimus); Arm D1 (TBI, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]; Arm D2 (busulfan, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]
Biological: Peripheral Blood Stem Cell — Given IV
  Other Names: PBSC; Peripheral Blood Stem Cells; peripheral stem cell; Peripheral Stem Cells
  Arms: Arm C1 (TBI, PTCy, tacrolimus); Arm C2 (busulfan, PTCy, tacrolimus); Arm D1 (TBI, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]; Arm D2 (busulfan, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]
Drug: Cyclosporine — Given IV
  Other Names: Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Cyclosporine Modified; Gengraf; Neoral; Sandimmune; SangCya
Drug: Sirolimus — Given IV
  Other Names: RAPA; Rapamune; rapamycin; SILA 9268A; WY-090217
Drug: Busulfan — Given IV
  Other Names: Bussulfam; Busulfanum; Busulphan; Busulfex; CB 2041; Glyzophrol; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: Arm A2 (busulfan, TnD); Arm C2 (busulfan, PTCy, tacrolimus); Arm D2 (busulfan, tacrolimus, methotrexate) [DISCONTINUED NOVEMBER 2021]
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration/biopsy
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase II trial investigates two strategies and how well they work for the reduction of graft versus host disease in patients with acute leukemia or MDS in remission. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms (Arms A and C).

ARM A: Patients are assigned to 1 of 2 arms.

ARM A1 (TBI BASED): Patients undergo total-body irradiation (TBI) twice daily (BID) on days -10 to -7, and receive thiotepa intravenously (IV) over 3 hours on days -6 and -5, fludarabine IV over 30 to 60 minutes on days -6 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, CD34+ enriched CD45RA-depleted donor T-lymphocytes IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

ARM A2 (BUSULFAN BASED): Patients receive fludarabine IV over 30 to 60 minutes on days -6 to -2, busulfan IV over 180 minutes on days -5 to -2, and undergo TBI BID on day -1. Patients also receive tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, CD34+ enriched CD45RA-depleted donor T-lymphocytes IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

ARM C: Patients are assigned to 1 of 2 arms.

ARM C1: Patients undergo TBI BID on days -4 to -2 or -3 to -1, and receive PBSC IV on day 0. Patients also receive cyclophosphamide IV over 1 to 2 hours on days 3 and 4, and tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day 5 approximately 24 hours after the end of the second dose of cyclophosphamide. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

ARM C2: Patients receive fludarabine IV over 30 to 60 minutes on days -5 to -2, busulfan IV over 180 minutes on days -5 to -2, PBSC IV on day 0, cyclophosphamide IV over 1 to 2 hours on days 3 and 4, and tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day 5 approximately 24 hours after the end of the second dose of cyclophosphamide. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

ARM D: (DISCONTINUED NOVEMBER 2021): Patients are assigned to 1 of 2 arms.

ARM D1: Patients undergo TBI BID on days -6 to -4, and receive cyclophosphamide IV over 1 hour on days -3 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, PBSC IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

ARM D2: Patients receive busulfan IV over 180 minutes on days -8 to -5, cyclophosphamide IV over 1 hour on days -3 to -2, tacrolimus (or cyclosporine or sirolimus if toxicities occur) IV continuously starting on day -1, PBSC IV on day 0, and methotrexate IV on days 1, 3, 6, and 11. If there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus (or cyclosporine or sirolimus) is tapered per month for capsules (or per week for liquid).

All patients also undergo bone marrow aspiration/biopsy, echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at days 7, 14, 21, 28, 56, 80, 180, and 270 and at 1, 1.5, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered appropriate candidates for myeloablative, TBI-containing allogeneic hematopoietic stem cell transplantation and have one of the following diagnoses:

  * Acute lymphocytic leukemia (ALL) in first or subsequent morphological remission (< 5% marrow blasts by morphology).
  * Acute myeloid leukemia (AML) in first or subsequent morphological remission (< 5% marrow blasts by morphology).
  * Other acute leukemia or related neoplasm (including but not limited to 'mixed phenotype' 'biphenotypic', 'acute undifferentiated' or 'ambiguous lineage' acute leukemia, blastic plasmacytoid dendritic cell neoplasm, lymphoblastic lymphoma, Burkitt leukemia/lymphoma, mast cell leukemia, chronic myeloid leukemia [CML] with blast crisis or other chronic myeloproliferative neoplasm) in first or subsequent morphological remission (<5% marrow blasts by morphology).
  * Myelodysplastic syndrome (MDS) with a history of excess blasts (≥ approximately 5% in marrow blasts by morphology) and a history of receiving cytoreductive therapy (including but not limited to BCL-2 inhibitors or cytotoxic chemotherapy) within the past 3 months.
* Patient age 1-60 years old (inclusive) at the time of informed consent

  * Patients aged 1-50 years old (inclusive) are eligible for TBI-based conditioning regimens.
  * Patients aged 1-60 years old (inclusive) are eligible for busulfan-based conditioning regimens (with or without TBI 4 Gy).
* Patient with an HLA-matched (HLA-A, B, C, DRB1, and DQB1 matched) related or unrelated donor capable of donating PBSC.
* Recipient informed consent/assent and/or legal guardian permission must be obtained.
* DONOR: HLA-matched related and unrelated donors (HLA-A, B, C, DRB1 and DQB1 matched based on high-resolution typing).
* DONOR: >= 18 years old.
* DONOR: Willing to donate PBSC.
* DONOR: Matched related donors:

  * Must give informed consent using the related donor informed consent form.
  * Must meet institutional donor eligibility criteria or be ineligible with statement that the donor is a first or second degree relative (exception 21 Code of Federal Regulations [CFR] 1271.65(b)(i)).
* DONOR: Matched unrelated donors:

  * Must consent according to the applicable National Marrow Donor Program (NMDP) donor regulatory requirements.
  * Must meet eligibility criteria as defined by the NMDP or be ineligible with statement of urgent medical need (exception 21 CFR 1271.65(b)(iii)).

Exclusion Criteria:

* Patients with central nervous system (CNS) involvement refractory to intrathecal chemotherapy and/or standard cranial-spinal radiation. A patient may have a history of CNS disease. However, any CNS disease must be cleared by the end of the pre-conditioning evaluation time frame. If CNS disease is identified on cerebrospinal fluid (CSF) evaluation within 30 days of the start of the preparative regimen a repeat CSF evaluation must be performed and show no evidence of disease in order for the patient to be eligible for the protocol.
* Patients on other experimental protocols for prevention of GVHD.
* Patient weight:

  * Patients with HLA-matched related donors will be excluded if they weigh >= 110 kg.
  * Patients with HLA-matched unrelated donors will be excluded if they weigh >= 110 kg and must be discussed with the Fred Hutch protocol principal investigator (PI) if they weigh >= 90 kg.
* Patients who are positive for human immunodeficiency virus (HIV)-1, HIV-2, human T-cell lymphotropic virus (HTLV)1 or HTLV2.
* Patients with uncontrolled infections for whom myeloablative HCT is considered contraindicated by the consulting infectious disease physician; i.e. patients with active infections require infectious disease consultation and documentation by the infectious disease team that myeloablative HCT is not considered to be contraindicated. Upper respiratory tract infection is not considered to represent an uncontrolled infection in this context.
* Patients with organ dysfunction, including:

  * Renal insufficiency (creatinine > 1.5 mg/dl) at the time of evaluation for the protocol. Patients with a known history of creatinine > 1.5 mg/dl or a current serum creatinine above the normal range for age must have a current creatinine clearance of > 60 ml/min/1.73 m^2 (measured by 24-hr urine specimen or nuclear glomerular filtration rate [GFR]).
  * Left ventricular ejection fraction < 45%.
  * Carbon monoxide diffusing capability (DLCO) corrected < 60%. Patients who are unable to perform pulmonary function tests (for example, due to young age and/or developmental status) will be excluded if the oxygen (O2) saturation is < 92% on room air.
  * Liver function abnormality. Patients who have liver function test (LFT)s (specifically, total bilirubin, aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) >= twice the upper limit of normal should be evaluated by a gastrointestinal (GI) physician unless there is a clear precipitating factor (such as an azole, MTX, trimethoprim-sulfamethoxazole, or another drug). If the GI physician considers that HCT on the protocol is contraindicated, that patient will be excluded from the protocol. Patients with Gilbert's syndrome require GI physician consultation but may be included on the protocol. Patients with no other known liver function abnormality or with reversible drug-related transaminitis do not necessarily require GI consultation and may be included on the protocol.
* Patients who have received previous myeloablative allogeneic or autologous transplantation.
* Patients with a life expectancy < 12 months from co-existing disease other than the leukemia or MDS.
* Patients who are pregnant or breast-feeding.
* Patients of childbearing age who are presumed to be fertile and are unwilling to use an effective birth control method or refrain from sexual intercourse during and for 12 months post-HCT.
* Patients with any other significant medical conditions that would make them unsuitable for transplantation, as determined by the PI.
* Patients with a known hypersensitivity to tacrolimus or MTX
* Patients who have received checkpoint inhibitors within three months of transplantation unless an exception is made by the PI
* DONOR: Donors who are HIV-1, HIV-2, HTLV-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection. Test must be performed using Food and Drug Administration (FDA) licensed, cleared, and approved test kits (serological and/or nucleic acid amplification test [NAT] and/or other approved testing) in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory.
* Unrelated donors donating outside of the USA.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Graft versus host disease (GVHD)-free relapse-free survival (RFS) | At 2 years
  Will be defined as survival-free of a history of: a) relapse after hematopoietic cell transplantation (HCT), b) grade III-IV acute GVHD after HCT, moderate or severe chronic GVHD meeting National Institutes of Health (NIH) criteria and requiring systemic pharmacologic immunosuppression for treatment of GVHD. RFS distribution will be estimated for each arm by the Kaplan-Meier curve, starting from the time of HCT. A 90% confidence interval (CI) will be constructed at 1 and 2-year post-HCT timepoints.

SECONDARY OUTCOMES:
Overall survival (OS) | At 2 years
  Death will be considered as the event, and the OS distribution will be estimated for each group by the Kaplan-Meier method, starting from the time of HCT. A 90% CI will be constructed at the 1 and 2-year post-HCT time points.
Relapse | At 2 years
  Will be defined as recurrence of leukemia (>= 5% leukemic blasts by flow or morphology) in bone marrow, circulating leukemic blasts or extramedullary disease (extramedullary disease definite i.e. proven by biopsy or probably based on clinical assessment if biopsy not feasible). Lower levels of leukemia in bone marrow or blood will be recorded and reported as 'measurable residual disease' but will not be considered relapse.
Proportion of patients alive and off prednisone (or equivalent systemic corticosteroid) for treatment of GVHD | At 3, 6, 9, 12, 15, 18, 21, 24 months post HCT
Graft rejection or irreversible graft failure (> 14 days duration) | At 2 years
  Will be operationally defined as failure to achieve an absolute neutrophil count (ANC) >= 0.5 x 10^9/L before death or second HCT, or decrease to ANC < 0.1 x 10^9/L for 14 consecutive days (date of graft failure defined as the 14th day) after an established donor graft despite daily administration of granulocyte colony-stimulating factor (subcutaneously or intravenously) and =< 20% bone marrow cellularity on bone marrow aspirate or biopsy any time in the first 2 years following HCT. If the delay or reduction in ANC is due to relapse (as determined by histopathology, flow cytometry or cytogenetic or molecular studies) this will not be considered graft failure. If a patient dies from organ toxicity and/or infection prior to day 28 without ANC >= 0.5 x 10^9/L this will not be considered graft failure.
Incidence of chronic GVHD | Up to 2 years
  Will be defined and graded based on NIH criteria and graded operationally as the occurrence of compatible symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bleakley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No